CLINICAL TRIAL: NCT03327714
Title: Mindfulness as a Method of Improving the Well-being, Quality of Life and Health of Primary School Pupils in Grades 0-9 (Ages 6-16)
Brief Title: Mindfulness as a Method of Improving the Well-being, Quality of Life and Health of Primary School Pupils
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016/299
Record Dates: First submitted 2017-09-29; First posted 2017-10-31 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Anxiety; Depression
Keywords: mindfulness; children; anxiety; depression; mental disorder; risk factor
MeSH Terms: conditions — Anxiety Disorders; Depression; Mental Disorders | interventions — Mindfulness

STUDY DESIGN:
Intervention Model Description: Children in classes that perform regular mindfulness are compared to children in classes that do not.

ARMS (2):
- Mindfulness and compassion (Experimental): Children aged between 6-16 years old will perform 5-10 minutes daily mindfulness and compassion training in school. The intervention will last for 10 weeks.
  Interventions: Behavioral: Mindfulness and compassion
- Control group (No Intervention): The control group consists of children who do not perform mindfulness in school.

INTERVENTIONS:
Behavioral: Mindfulness and compassion
  Arms: Mindfulness and compassion

SUMMARY:
This study evaluates the short and long-term effect of 5-10 minutes daily mindfulness and compassion training in school among children aged between 6-16 years old. The mindfulness intervention will last for 10 weeks and the results will be compared to children who do not perform mindfulness in school. Due to practical reasons, the study is not randomized; classes are instead placed in the mindfulness or control group. Anxiety, mental, physical and social health, quality of life, and school performance will be evaluated via questionnaires and school registries, before and after the intervention and thereafter once a year until the end of ninth grade (age 16 years). Long term health (diagnoses, medical consumption, and drug prescriptions) and family income (proxy for socioeconomic status) will be followed in regional and national registries until 25 years of age.

The hypothesis of the study is that mindfulness can prevent mental disorders and anxiety, and increase well-being in children and adolescents. The primary aim is to subsequently evaluate if regular, daily, mindfulness and compassion training (5-10 minutes) prevents anxiety and mental disorders in children and adolescents. Secondary aims are to evaluate 1) the effect of mindfulness on daily life, quality of life, and health in school pupils; 2) the effect of mindfulness on school performance; 3) the effect of mindfulness and compassion on the class room environment; 4) the effect of potential individual, family, and school-level risk factors on mental health in children and adolescents; 5) the effect of mindfulness on these potential risk factors.

Sessions are led by school teachers who have been educated in mindfulness. Their own levels of stress and mindfulness will be evaluated by a questionnaire and compared to teachers in control classes both before and after the intervention. The teachers will also be interviewed to evaluate the effect of mindfulness on the class room environment.

In a sub-study, the effect of mindfulness on brain structure and function will be examined by magnetic resonance imaging in school pupils aged 15-16 year old. This will be preceded by a pilot study, in which feasibility of the method is tested in the target group.

To achieve sufficient statistical power, taking into account a cluster effect to adjust for grouping of the pupils, 1750 children and adolescents will be recruited. Written informed consent is a prerequisite for participation.

ELIGIBILITY:
Inclusion Criteria:

* School pupils in grade 0-9

Exclusion Criteria:

* No exclusion criteria

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1750 (Estimated)
Dates: Start 2016-10-12 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2039-06-30 (Estimated)

PRIMARY OUTCOMES:
Effect of mindfulness on change in anxiety and depression in children, grade 3-9, as measured by the Beck Depression Inventory for Youth and the Beck Anxiety Inventory for Youth. | Change from baseline depression and anxiety levels at 10 weeks
  The primary aim is to evaluate if regular, daily, mindfulness and compassion practice (5-10 minutes) for 10 weeks prevents anxiety and depression in children, grade 3-9. Results will be compared within respective group (change from baseline) and between mindfulness and control group.

SECONDARY OUTCOMES:
Effect of mindfulness on changes in daily life as measured by questions about school and leisure time (adapted from the Scania Public Health Survey). | Change from baseline daily life status at 10 weeks
  To evaluate the effect of regular mindfulness on daily life in children, grade 0-9, as measured by a number of questions about school and leisure time (adapted from the Scania Public Health Survey).
Effect of regular mindfulness practice on school performance (data collected from school registers) | Grade 0 (pupils aged 6-7 years) and will continue on a yearly basis until grade 9 (pupils aged 15-16).
  To evaluate the effect of regular mindfulness on grades and attendance. The report cards will be collected before the Swedish summer holidays commence in June
Effect of mindfulness on change in class room environment (evaluated by questionnaires, weekly schedule, and interviews with teachers). | Change from baseline class room environment at 10 weeks
  To evaluate the effect of regular mindfulness on class room environment (evaluated by questionnaires, weekly schedule, and interviews with teachers).
Effect of risk factors on mental health: longitudinal follow-up study. | Baseline, 10 weeks, 52 weeks. Thereafter yearly until 25 years of age.
  To evaluate the association between, and effect of, potential individual, family, and school-level factors on mental health in children and adolescents. First results are obtained at baseline via questionnaires, the next 10 weeks later. Thereafter yearly until ninth grade (questionnaires) and until 25 years of age (diagnoses via registers)
Effect of mindfulness on risk factors: longitudinal follow-up study. | 10 weeks, 52 weeks. Thereafter yearly until 25 years of age.
  The effect of mindfulness on potential individual, family, and school-level risk factors. First evaluation after 10 weeks. Thereafter yearly until ninth grade (questionnaires) and 25 years of age (diagnoses via registers).
Effect of mindfulness on changes in quality of life as measured by questions adapted from the Scania Public Health Survey and Living Conditions Surveys (ULF/SILC) | Change from baseline quality of life at 10 weeks
  To evaluate the effect of regular mindfulness on quality of life in children, grade 0-9, as measured by questions adapted from the Scania Public Health Survey and Living Conditions Surveys (ULF/SILC)
Effect of mindfulness on changes in health as measured by questions about school and leisure time (adapted from the Scania Public Health Survey). | Change from baseline health at 10 weeks
  To evaluate the effect of regular mindfulness on health in children, grade 0-9, as measured by a number of questions about general health (adapted from the Scania Public Health Survey)
Long-term effect of mindfulness practice on anxiety, depression, daily life, quality of life and health as measured by the BDI Youth, the Scania Public Health Survey and Living Conditions Surveys (ULF/SILC) and registries: longitudinal follow-up study | 52 weeks and thereafter yearly until 25 years of age.
  Long-term follow-up of outcomes # 1, 2, 7 and 8 via questionnaires once a year until ninth grade, and health until 25 years of age (diagnoses via registers)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Sundquist, PhD, MD, Principal Investigator — Center for Primary Health Care Research, Institution of Clinical Sciences, Malmö, Sweden
Locations (1):
- Center for Primary Health Care Research, Malmo, Sweden